CLINICAL TRIAL: NCT03689660
Title: The Feasibility of Virtual Reality in Children With Neuromuscular Disease and the Effectiveness of Virtual Reality and Biofeedback Training on Functional Levels of Children With Neuromuscular Disease
Brief Title: Feasibility of Virtual Reality in Children With Neuromuscular Disease, Effectiveness of Virtual Reality and Biofeedback
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Merve Kurt (Other)
Responsible Party: Sponsor-Investigator, Merve Kurt, Research Assistant, Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Merve Kurt
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Neuromuscular Disease; Duchenne Muscular Dystrophy; Spinal Muscular Atrophy; Virtual Reality; Biofeedback
Keywords: motivation; neuromuscular disease; duchenne muscular dystrophy; spinal Muscular Atrophy; virtual reality; biofeedback training
MeSH Terms: conditions — Neuromuscular Diseases; Muscular Dystrophy, Duchenne; Muscular Atrophy, Spinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Nope
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Training (Experimental): Virtual reality treatment will be applied during the 12 weeks. The training will consist of three sessions per week and 30 minutes per session.
  Interventions: Other: Virtual Reality Training
- Biofeedback Training (Experimental): Biofeedback training will be applied during the 12 weeks. The training will consist of three sessions per week and 30 minutes per session.
  Interventions: Other: Biofeedback Training
- Conventional Rehabilitation (Other): Participants will continue this rehabilitation program if they are already getting rehabilitation in a rehabilitation center. If they do not participate in any rehabilitation program, they will be included in the conventional rehabilitation program by us.
  Interventions: Other: Conventional rehabilitation

INTERVENTIONS:
Other: Virtual Reality Training — Participants will be given a game-based workout program that includes balance and weight transfers using the XBOX Kinect ™ device in a low-to-medium intensity for 3 weeks, 3 days a week, 30 minutes per day.
  Arms: Virtual Reality Training
Other: Biofeedback Training — biofeedback training will be applied to participants in 10-minute sessions with 10 seconds of voluntary contraction and 15 seconds of rest at each session. Training will last 12 weeks.
  Arms: Biofeedback Training
Other: Conventional rehabilitation — Participants will receive a 12-week conventional rehabilitation program.
  Arms: Conventional Rehabilitation

SUMMARY:
Our study is a randomized controlled study and the subjects included in the study will be divided into three groups as virtual reality training, biofeedback training, and conventional rehabilitation.

DETAILED DESCRIPTION:
We have 3 purposes:

1. Determine the feasibility of virtual reality training in children with neuromuscular disease.
2. To determine the effect of virtual reality, biofeedback training, and conventional rehabilitation on functional levels and balances of children with neuromuscular disease.
3. To compare the motivation of children with neuromuscular disease to virtual reality, biofeedback training, and conventional rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study
* Being diagnosed with the neuromuscular disease
* No other systemic or neurological disease
* No significant visual or auditory loss
* Continuation of ambulation (10 m walking independently)
* Be able to understand simple commands

Exclusion Criteria:

* Performing a drug change at 3 months before treatment or during treatment which may affect muscle strength
* Acute inflammation in the musculoskeletal system
* Finding any orthopedic problem that prevents activities during the research

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
The Motor Function Measure-32 | 30 minutes
  MFM-32 is a scale developed to evaluate motor functions of children and adults with neuromuscular disease. The scale can be used to evaluate both in children with and without walking problems.The MFM-32 consists of 32 items. Each item is answered with a 4-point likert scale (0 = cannot initiate the exercise or maintain its starting position, 1 = partially completes the exercise, 2 = completes exercises with compensations, slowly or roughly, 3 = completes the exercise in the standard pattern). The scale can be used for the evaluation of individuals aged between 6 and 60 years.
Pediatric Functional Independence Measure | 5 minutes
  WeeFIM consists of 18 items divided into 6 sub-scales (self-care, sphincter control, mobility, locomotion, communication, social communication). Each item is scored from 1 to 7. A higher score indicates a better functional level.
Balance Master System | 20 minutes
  The static and dynamic balance evaluated using the Balance Master System ver. 8.1. (NeuroCom International Inc. Clackamas, OR, USA) force platform system which has multiple testing protocols designed to examine balance. The system includes a computer linked force plate that records data with the aid of crystal transducers.
Vignos Scale | 2 Minutes
  The Vignos Scale has been developed to evaluate the lower extremity functions. The scale allows the lower extremity functions to be scored between 1 (can walk and climb stairs without help) and -10 (bed dependent).
Feasibility of Virtual Reality | 1 Minutes
  The feasibility of virtual reality will be examined by laboratory tests. Laboratory tests to be carried out are as follows: Creatine Kinase, Lactate Dehydrogenase (LDH), Myoglobin, Serum Electrolytes, C-Reactive Protein levels. These are agents that are indicative of muscle destruction or inflammation. Will be evaluated in order to follow muscle destruction.
Pediatric Motivation Scale | 5 Minutes
  The PMOT is recommended for assessing motivation to rehabilitation program in children aged 8 to 18 years. It comprises six subscales (effort-importance, interest-enjoyment, competence, relatedness, autonomy, and value-usefulness) with total 21 items. While the 19 items of the scale are answered with a 6-point smiley face scale (1 = absolutely false, 6 = absolutely correct), there are 2 open-ended questions on the scale. The high scores in each sub-scales indicate that the child's motivation in that sub-section is high. A higher total score indicates that the motivation is intrinsically arranged and that the child has a high motivation. From this point of view, the scale gives information about both the type of motivation and the amount of motivation of the child.
Visual Analog Scale | 1 Minute
  Visual Analog Scale will be applied to evaluate muscle pain. It has a fixed line between two end adjectives of 100 mm length. The end adjectives in our study will be "no pain" and "too much pain".

SECONDARY OUTCOMES:
Pediatric Functional Reaching Test | 1 Minute
  For the Pediatric Functional Reach test, children will be asked to raise their arms 90o in an upright posture position, extending to the maximum possible distance in three directions, forward, right, and left. Reach distances will be measured by pointing the wall with the end point of the third finger, and distances; "start", "final" and "difference" will be determined in cm using tape measure.
Fall Frequency | 1 Minute
  The frequency of the fall will be questioned with a chart created by the researchers. The family will be asked to record the children's each fall a week before the study and a week after the treatment.
Muscle Strength Test with Hand Held Dinamometer | 20 minutes
  Upper and lower limb muscles strength will be evaluated with hand held dinamometer device. This device allows recording of muscle strength in kilograms.
Timed Up Go Test | 2 Minutes
  For the time up go test, children will be asked to walk with two walking cones at a distance of 10 meters, at normal walking speeds, and the elapsed time will be recorded in seconds.
Stair Climb Test | 2 Minutes
  Children will be asked to climb up and down as quickly as they can, without running the steps, on a ladder of 16-20 cm height and 8-14 steps and the elapsed time will be recorded in seconds.
T-shirt Wear Remove Test | 2 Minutes
  For the T-shirt pull-out test, the children will be asked to wear a T-Shirt in the sitting position as soon as possible and the elapsed time will be recorded in seconds; then they will be asked to remove the T-Shirt as soon as possible and the elapsed time will be recorded in seconds.
Stand Up from Supine Position Test | 1 Minutes
  From the supine position to stand up, children will be asked to lie on the back of the body, the arms next to the body, the legs as closed as possible, and the head on the midline on a mat. Then, from this position, they will be asked to stand as soon as possible and the elapsed time will be recorded in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Tülay Tarsuslu Şimşek, Study Director — Professor Dr.
Locations (1):
- Dokuz Eylul University, Izmir, Balcova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The IPD may share when requested
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD: Balance results, Functional Level, Diagnosis, demographic data
Access Criteria: The IPD may share when requested.